CLINICAL TRIAL: NCT05456880
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of a Single Dose of Autologous CD34+ Base Edited Hematopoietic Stem Cells (BEAM-101) in Patients With Sickle Cell Disease and Severe Vaso-Occlusive Crises (Beacon Trial)
Brief Title: BEACON: A Study Evaluating the Safety and Efficacy of BEAM-101 in Patients With Severe Sickle Cell Disease
Acronym: BEACON
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTX-AUT-001
Record Dates: First submitted 2022-06-23; First posted 2022-07-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Gene Editing; Sickle Cell; Severe Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BEAM-101 (Experimental): BEAM-101 manufactured with autologous CD34+ hematopoietic stem cells collected by plerixafor mobilization and edited ex vivo. No maximum dose has been set for BEAM-101; all of the gene edited cells that pass release specifications will be administered to the patient. BEAM 101 will be administered as a single dose by IV infusion.
  Interventions: Biological: BEAM-101

INTERVENTIONS:
Biological: BEAM-101 — Single dose of BEAM-101 administered by IV following myeloablative conditioning with busulfan

SUMMARY:
This is an open-label, single-arm, multicenter, Phase 1/2 study evaluating the safety and efficacy of the administration of autologous base edited CD34+ HSPCs (BEAM-101) in patients with severe SCD

ELIGIBILITY:
Key Inclusion Criteria Include:

1. Age ≥12 years to ≤35 years
2. Documented diagnosis of sickle cell disease with βS/βS, βS/β0, or βS/β+ genotypes.
3. Severe SCD defined by the occurrence of at least 4 severe VOCs in the 24 months prior to screening despite receiving hydroxyurea or other supportive care measures

Key Exclusion Criteria Include:

1. HbF levels >20%, obtained at the time of screening on or off hydroxyurea therapy
2. Previous receipt of an autologous or allogeneic HSCT or solid organ transplantation
3. Available and willing matched sibling donor
4. Definitive diagnosis of moyamoya syndrome based on screening brain MRA
5. History of overt stroke

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in annualized number of severe VOCs (Vascular-occlusive Crisis) relative to baseline | 6 months to time of analysis as compared to baseline
Proportion of patients with successful neutrophil engraftment | BEAM-101 administration to month 24
Time to neutrophil engraftment | BEAM-101 administration to month 24
Time to platelet engraftment | BEAM-101 administration to month 24
Transplant-related mortality within 100 days after beam-101 treatment | BEAM-101 administration to day 100
Safety and tolerability assessments based on frequency, severity and seriousness of adverse events (AE's) | BEAM-101 administration through month 24

SECONDARY OUTCOMES:
Proportion of patients experiencing at least 75% reduction in annualized rate of severe VOCs | Month 6 post BEAM-101 treatment to month 24 as compared to baseline
Proportion of patients experiencing no severe VOCs | 6 months to time of analysis as compared to baseline
Change in annualized number of hospitalizations for VOCs | Month 6 post BEAM-101 treatment to month 24 as compared to baseline
Change in annualized duration of hospitalizations for VOCs | Month 6 post BEAM-101 treatment to month 24 as compared to baseline
Change in RBC transfusions per month and per year for SCD-related indications | Month 2 post BEAM-101 treatment to month 24 as compared to baseline
Change in total Hgb (g/dL) concentration over time | Baseline to month 24
Proportion of patients with HbF ≥30%, for at least 3 months | Month 6 post BEAM-101 treatment to month 24 as compared to baseline
Change in lactate dehydrogenase (LDH) over time | Month 3 post BEAM-101 treatment to month 24 as compared to baseline
Change in total bilirubin over time | Month 3 post BEAM-101 treatment to month 24 as compared to baseline
Change in free Hgb over time | Month 3 post BEAM-101 treatment to month 24 as compared to baseline
Change in haptoglobin over time | Month 3 post BEAM-101 treatment to month 24 as compared to baseline
Change in reticulocyte count over time | Month 3 post BEAM-101 treatment to month 24 as compared to baseline

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta - Aflac Cancer and Blood Disorders Center - Egleston Hospital, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Henry Ford Cancer Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ligon JA, Cupit-Link MC, Yu C, Levine J, Foley T, Rotz S, Sharma A, Gomez-Lobo V, Shah NN. Pediatric Cancer Immunotherapy and Potential for Impact on Fertility: A Need for Evidence-Based Guidance. Transplant Cell Ther. 2024 Aug;30(8):737-749. doi: 10.1016/j.jtct.2024.06.006. Epub 2024 Jun 10. PMID 38866240
- [Derived] Sharma A, Young A, Carroll Y, Darji H, Li Y, Mandrell BN, Nelson MN, Owens CL, Irvine M, Caples M, Jerkins LP, Unguru Y, Hankins JS, Johnson LM. Gene therapy in sickle cell disease: Attitudes and informational needs of patients and caregivers. Pediatr Blood Cancer. 2023 Jun;70(6):e30319. doi: 10.1002/pbc.30319. Epub 2023 Mar 28. PMID 36975201
- [Derived] Persaud Y, Mandrell BN, Sharma A, Carroll Y, Irvine M, Olufadi Y, Kang G, Hijano DR, Rai P, Hankins JS, Johnson LM. Attitudes toward COVID-19 vaccine among pediatric patients with sickle cell disease and their caregivers. Pediatr Blood Cancer. 2023 May;70(5):e30274. doi: 10.1002/pbc.30274. Epub 2023 Mar 1. PMID 36860093